CLINICAL TRIAL: NCT00278239
Title: Study of Outcome of Children Previously Enrolled in European Trials of Treatment for Primitive Neuroectodermal Tumour (PNET)
Brief Title: Quality of Life in Patients Who Have Undergone Previous Treatment for Primitive Neuroectodermal Tumors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000454509; CCLG-CNS-2002-03; EU-20578
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2006-04

CONDITIONS: Brain and Central Nervous System Tumors; Cognitive/Functional Effects; Long-term Effects Secondary to Cancer Therapy in Children; Psychosocial Effects of Cancer and Its Treatment
Keywords: long-term effects secondary to cancer therapy in children; psychosocial effects of cancer and its treatment; cognitive/functional effects; childhood supratentorial primitive neuroectodermal tumor
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Mental Status and Dementia Tests; Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: cognitive assessment
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Questionnaires that measure quality of life may improve the ability to plan treatment for patients with primitive neuroectodermal tumors.

PURPOSE: This phase III trial is studying quality of life in patients who have undergone previous treatment for primitive neuroectodermal tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the quality of survival of patients in the UK and other European countries enrolled in previous International Society of Pediatric Oncology (SIOP) 2 or 3 phase III trials for treatment of pediatric primitive neuroectodermal tumors (PNET).
* Compare the quality of survival between children allocated to different treatments in these trials.

Secondary

* Determine the framework that will allow similar information to be collected across all participating countries in the PNET 4 trial that opened in autumn 2002.

OUTLINE: This is a cross-sectional, multicenter study.

Pediatric oncologists, teachers, patients ≥ 12 years old, and parents of children age 3-11 years old complete six questionnaires to assess the patients' motor and sensory function, cognition, behavior, emotion, educational provision and achievement, social integration, and the subjective experience of the patients and their families.

PROJECTED ACCRUAL: A total of 229 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Surviving primitive neuroectodermal tumor (PNET) patients previously enrolled in International Pediatric Oncology Society (SIOP) 2 or 3 phase III treatment trials
* Surviving PNET patients eligible for and treated according to PNET 3 protocol but not randomized
* No metastatic disease at time of allocation to treatment
* No current progressive disease

PATIENT CHARACTERISTICS:

* No patient deemed unsuitable for this study by treating clinician

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 3 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2002-06

PRIMARY OUTCOMES:
Quality of life (QOL) as measured by QOL questionnaire

SECONDARY OUTCOMES:
Quality of survival compared among children undergoing different treatments by Health Utilities Index

CONTACTS AND LOCATIONS:
Overall Officials: Colin Kennedy, Study Chair — University Hospital Southampton NHS Foundation Trust
Locations (21):
- Our Lady's Hospital for Sick Children, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children NHS Trust, London, England
  - Central Manchester and Manchester Children's University Hospitals NHS Trust, Manchester, England
  - Sir James Spence Institute of Child Health, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales